CLINICAL TRIAL: NCT05091957
Title: CONNECTING FAMILIES: A Randomized Controlled Trial of Primary Care Poverty Screening and Financial Support Navigation for Families of Young Children
Brief Title: Connecting Families
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Imaan Bayoumi, Associate Professor, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: FMED-6797-21
Record Dates: First submitted 2021-09-14; First posted 2021-10-25 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Poverty; Primary Care; Intervention

STUDY DESIGN:
Intervention Model Description: A multi-centred, pragmatic, 1:1 allocation, parallel-group superiority randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Community Support Worker (Experimental): structured review of participant income supports with a trained CSW, to identify financial needs and benefits for which the family is eligible, including assessment of income and food security, affordability of medications, housing and energy insecurity, and dental care. The visits will be conducted in person, by telephone or by videoconferencing, according to participant preference and to ensure adherence to COVID-19 pandemic-related criteria.
  Interventions: Other: Community Support Worker
- Usual Care (Active Comparator): There is no clear standard of care and potential for practice variation in clinician responses to identified social need. Based on the ethical imperative to provide some support to families who identify unmet social needs, the comparator group will receive Usual Care, defined as: Participants in both groups will receive a written summary of available resources.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Community Support Worker — structured review of participant income supports with a trained CSW, to identify financial needs and benefits for which the family is eligible, including assessment of income and food security, affordability of medications, housing and energy insecurity, and dental care. The visits will be conducted in person, by telephone or by videoconferencing, according to participant preference and to ensure adherence to COVID-19 pandemic-related criteria.
  Arms: Community Support Worker
Other: Usual Care — Participants in both groups will receive a written summary of available resources
  Arms: Usual Care

SUMMARY:
Living in poverty has a profound negative impact on parenting stress and children's health. When poverty occurs early in childhood and continues for a long time, the impact on child health can be lifelong. Child poverty is common, affecting about 20% of Canadian children. Many low income families may not be receiving all the social benefits for which they are eligible. There are calls for primary care providers to ask patients if they have difficulty making ends meet at the end of the month and to intervene if poverty is identified, but it is not known if intervening can improve parent's and children's health. This study will test whether a Community Support Worker who helps families with young children navigate the social service system by reviewing social needs (like food, housing or energy insecurity) and income supports can lead to increased family income, reduced parenting stress and an improvement in their child's health. The Community Support Worker will help families complete income tax, apply for benefits and community supports for which they are eligible. The investigators will also study the effect of this intervention on health care utilization. Our study will be conducted in Toronto and Kingston in primary care practices participating in the TARGet Kids! primary care research network. Results from this study will help health care providers and policy makers understand whether Community Support Workers are an effective way to integrate the health and social service systems to improve parent and child health.

DETAILED DESCRIPTION:
INTRODUCTION AND IMPORTANCE: Poverty and financial strain have profound and long-lasting negative impacts on both parent and child health, contributing to substantial health disparities. As the first contact with the health system for most families, primary care providers are uniquely positioned to address child poverty in clinical settings.

Many professional health organizations recommend that healthcare providers identify and address social determinants of health, but there is little evidence regarding the impact of effective interventions. Social systems are frequently complex and difficult to navigate; for example, low income Canadians are known to have lower tax filing rates than the general population. Therefore, many families may not be accessing all social benefits to which they are entitled. The investigators propose to rigorously test a poverty reduction intervention (navigation of financial supports) embedded in primary care using a randomized controlled trial to evaluate the impact on parent and child health outcomes. Results of our pilot study demonstrated feasibility and will inform our proposed full trial.

METHODS: Study Design: A multi-site, pragmatic, blinded, superiority, parallel-group randomized controlled trial will be conducted.

Participants: Families of children ages (from birth to 2 years), screening positive for the question "Do you ever have difficulty making ends meet at the end of the month?", identified as a good predictor of poverty.

Intervention and Active Comparator: Families will be randomly allocated to the intervention or active comparator group. Parents in the intervention group will have a review of their social needs and resources with a trained Community Service Worker (CSW) with a thorough understanding of potential income supports and community agencies and will assist the parent to access financially related social benefits for which they are eligible. All participants will receive a written summary of available resources.

Outcomes: The primary outcome, measured 6 months after enrollment, is parenting stress, as measured by the Parenting Stress Index-Short Form. Secondary outcomes are change in: a) self-reported after-tax household income; b) household food security; c) parent depression; d) child development; e) child social, emotional and behavioural health; f) Community Service Worker workload; g) health care utilization.

TEAM EXPERTISE: The study is a collaboration between TARGet Kids!, (a well-established child-focused primary care practice-based research network) and integrated Knowledge Users (parents, administrators and policy makers). The research team has expertise in child health, pragmatic trials and social determinants of health.

EXPECTED OUTCOME: Results from this research will address a critical evidence gap regarding a feasible and scalable intervention to address child poverty in the primary care practice setting. Leveraging primary preventive care in early childhood, which is accessed by almost all families, will provide powerful opportunities for implementation. Effective interventions to address child poverty and financial strain in clinical practice have the potential to influence child health trajectories over their life course.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children (younger than 3 years) attending a regularly scheduled primary care visit.
* Parents respond affirmatively to the question "Do you ever have difficulty making ends meet at the end of the month?"
* Informed parental consent. Only one child will be enrolled per family. For families with more than one child, we will enroll the youngest eligible child, since literature suggests that impact of reducing family stress may be greater at younger ages; for multiple births, one child will be randomly selected for inclusion.

Exclusion Criteria:

1. Parents without legal status in Canada, as they are not eligible for many Canadian social programs.
2. Families who are receiving system navigation support, such as from a social worker or public health nurse, or who have received system navigation support within one year prior to enrolment.
3. Child with a previously diagnosed developmental disorder, genetic, chromosomal or syndromic condition.
4. Child born prematurely (gestational age less than 32 weeks).

Ages: 1 Day to 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Self reported
Enrollment: 80 (Estimated)
Dates: Start 2022-05-17 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Parenting Stress Index- Short Form 4 | 6 months
  A 36-item parent-completed questionnaire assessing overall level of stress a person is feeling in their role as a parent. Scoring yields an overall stress score (range 36-180, with higher scores indicating greater stress) and sub-scores for Parental Distress, Parent-Child Dysfunctional Interaction and Difficult Child (each with range of 5-60) which are summed to generate the total score. .

SECONDARY OUTCOMES:
Self Reported Household Income | 6 months, 12 months
  Self Reported Household Income from all sources
Participant use of community resources | 6 months, 12 months
  This is a study specific instrument which assesses participants' receipt of a comprehensive suite of financial benefits (including specific income tax benefits, benefits through social assistance programs) and receipt of emergency food services, childcare subsidy, energy assistance, support for medication and dental costs and housing needs.
Household food security | 6 months, 12 months
  18-item Household Food Security Survey Module, asks about the household's experiences of food insecurity during the previous year. Higher scores indicate increased food insecurity and households are classified as food secure, marginally food insecure, moderately food insecure or severely food insecure.
Social Needs | 6 months, 12 months
  WE Care Survey, s a 10-item questionnaire assessing needs in 4 domains (economic stability, education, neighborhood & physical environment, and food) and whether participants want help with identified needs..
Parent Depression | 6 months, 12 months
  Patient Health Questionnaire - 9, a 9 item self completed instrument measuring symptoms of depression (range 0-27 with higher scores indicating worse outcome).
Parent anxiety | 6 months, 12 months
  Generalized Anxiety Disorders-7, a 7 item self completed instrument measuring symptoms of anxiety (range 0-21, with higher scores indicating worse outcome).
Child Social- Emotional Development | 6 months,12 months
  Ages and Stages: Social Emotional, age specific parent completed questionnaires assessing the child's social and emotional development, in which higher scores indicate better outcomes.
Child general development | 6 months, 12 months
  Ages and Stages-3: age specific parent completed questionnaires assessing the child's s development in 5 developmental areas (Communication, Gross Motor, Fine Motor, Problem Solving, Personal Social), in which higher scores indicate better outcomes.
Pediatric health system utilization | 6 months, 12 months
  Through linkage with health administrative databases, the investigators will assess differences in health services utilization. The following administrative databases will be used: Ontario Health Insurance Plan (OHIP) which includes physician billings (fee for service and shadow billing) for physician visits, the National Ambulatory Care Reporting System (NACRS) which includes data on emergency department visits, and the Discharge Abstracts Database (DAD) which includes data on inpatient hospitalizations. We will assess between-group differences in primary care visits, low acuity emergency department visits (CTAS 3-5), number of hospitalizations and length of stay.For children, primary care visits will be categorized as well-child visits (which may appropriately increase) and other visits (which may be reduced).
Parent health system utilization | 6 months, 12 months
  Through linkage with health administrative databases, the investigators will assess differences in health services utilization. The following administrative databases will be used: Ontario Health Insurance Plan (OHIP) which includes physician billings (fee for service and shadow billing) for physician visits, the National Ambulatory Care Reporting System (NACRS) which includes data on emergency department visits, and the Discharge Abstracts Database (DAD) which includes data on inpatient hospitalizations.We will assess between-group differences in primary care visits, low acuity emergency department visits (CTAS 3-5), number of hospitalizations and length of stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's Family Health Team, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
All deidentified data relevant to the study will be made available upon reasonable request to the principal investigators.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning with publication of main study results to 5 years later.
Access Criteria: Upon reasonable request directed to the principal investigators via email.

REFERENCES:
- [Derived] Bayoumi I, Parkin PC, Tabassum F, Johnson C, Sherwood M, Mitchell M, Birken CS, Bloch G, Carsley S, Cole M, Green M, Keown-Stoneman CDG, Maguire JL, Purkey E, van den Heuvel M, Weir S, Wong P, Borkhoff CM. Connecting families-randomised controlled trial of poverty screening and financial support navigation for families of young children in primary care: an internal pilot study informed protocol. BMJ Open. 2026 Feb 6;16(2):e111158. doi: 10.1136/bmjopen-2025-111158. PMID 41651520